CLINICAL TRIAL: NCT06652581
Title: Effectiveness Of Modified-Thoracoabdominal Nerve Block Perichondrial Approach (M-TAPA) Post-Operative Analgesia Compared To Intravenous Opioids In Laparoscopic Cholecystectomy Patients
Brief Title: Effectiveness Of Modified-Thoracoabdominal Nerve Block Perichondrial Approach (M-TAPA) In Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, amelia christiana, Principle Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2176/UN14.2.2.VII.14/LT/2024
Record Dates: First submitted 2024-10-01; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Laparoscopic Cholecystectomy; Peripheral Nerve Block
Keywords: Analgesia; Laparoscopy Cholecystectomy; Peripheral Nerve Block; Pain management; Ultrasound; Postoperative Pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Thorachoabdominal Nerve Block Perichondrial Approach(M-TAPA) (Experimental): USG Guided Bilateral Modified Thorachoabdominal Nerve Block Perichondrial Approach (M-TAPA) using 20 ml Bupivacaine 0,25%.
  Interventions: Procedure: Modified Thorachoabdominal Nerve Block Perichondrial Approach(M-TAPA
- Opioid Intravena (Active Comparator): This Group receive opioid intravena post surgery without M-TAPA Block
  Interventions: Device: Opioid Intravena

INTERVENTIONS:
Procedure: Modified Thorachoabdominal Nerve Block Perichondrial Approach(M-TAPA — USG Guided Bilateral Modified Thorachoabdominal Nerve Block Perichondrial Approach (M-TAPA) using 20 ml Bupivacaine 0,25%.
  Other Names: P1
  Arms: Modified Thorachoabdominal Nerve Block Perichondrial Approach(M-TAPA)
Device: Opioid Intravena — Opioid Intravenous post Surgery without M-TAPA Block delivered with PCA Machine
  Other Names: P2
  Arms: Opioid Intravena

SUMMARY:
The Goal of this clinical trial is to determine the advantages of using Peripheral Nerve Block by injecting drugs under the skin on both sides of the abdomen in the upper abdominal area in patients undergoing laparoscopic Cholecystectomy. Study participants will be divided into 2 groups, namely group P1 receiving Modified Thoracoabdominal Perichondrial Approach (M-TAPA) block anesthesia after laparoscopic cholecystectomy and group P2 only receiving intravenous opioids postoperatively. Peripheral nerve blocks on both sides of the upper abdomen are expected to be able to prolong the duration of pain relief, reduce the pain scale, and the total dose of pain medication needed postoperatively. The injection of this peripheral nerve block drug will be carried out by an anesthesiologist. Researchers will continue to anticipate the occurrence of side effects that can occur with strict monitoring and emergency care standards. This study will last up to 24 hours after surgery.

The main question it aims to answer is:

To prove that the amount of postoperative intravenous opioid consumption with M-TAPA block is lower than the control group.

DETAILED DESCRIPTION:
A. Treatment of patients in P1 and P2 before entering the operating room:

1. Every patient who meets the eligibility criteria will be asked for consent to become a subject of this study. Proof of consent is the signing of a letter of willingness to become a subject of the study by the informant, the consent giver, and one witness. Quality of Recovery using QoR 40 form will evaluate before surgery and 24 hours after surgery.
2. Patients have been fasted for 8 hours from solid food before surgery, clear water up to 2 hours before surgery. The infusion is installed 2 hours before the patient is sent to the operating room using an 18G intravenous catheter with Ringer lactate fluid at a rate of administration according to the patient weight 10 ml/kg/hour

B. Treatment of patients in the operating room P1 and P2:

1. General anesthesia was performed in both groups.
2. General anesthesia begins with preoxygenation for 3-5 minutes with 100% O2.
3. Continued induction using intravenous propofol 2 mg/kgBW and intravenous fentanyl 2 mcg/kgBW.
4. After the patient is induced, continue by giving the muscle relaxant atracurium 0.5 mg/kgBW intravenously.
5. After three minutes, laryngoscopy and intubation are performed using an endotracheal tube (ETT) with a size according to the patient needs.
6. Maintain anesthesia with oxygen and compressed air with a ratio of 1 liter: 1 liter and sevoflurane.
7. All patients were performed with the same laparoscopic cholecystectomy procedure (4-port technique), umbilical port (5mm), infraxiphoidal (15-20 mm), lateral intersection of the umbilicus and axillary line (5 mm), and symmetrical assistant port (5 mm). With a pneumoperitoneum pressure of 10-12 mmHg.
8. Continue with the operation until completion. One hour before the surgery is completed, the patient is given anti-vomiting prophylaxis ondansetron 0.1 mg/kgBW intravenously.

Group P1:

1. Continue with preparation for the block procedure on the patient.
2. After the necessary tools and materials are ready, the Anesthesiologist who will perform the block washes his hands sterilely, uses a sterile gown and gloves.
3. Then the area of action is disinfected, with the sequence of 70% alcohol, betadine, 70% alcohol then a sterile hole drape is installed.
4. Identification of the place to perform the block is carried out, namely between the midclavicular line and the anterior axillary. The injection identification guide uses ultrasound.
5. The ultrasound machine uses a linear probe placed on the chondrium with a sagittal cut at Costa 10, identifying the external oblique muscle, internal oblique, transversus abdominis, costal cartilage. Stimuplex 22Gx50mm is injected using the in-plane technique. The tip of the needle is placed under the chondrium.
6. Before injecting local anesthetic drugs, negative aspiration (exclusion of intravascular injection) and hydrodissection using 0.9% NaCl as much as 1 - 2 ml are performed to further ensure the area of the needle tip. Local anesthetic bupivacaine 0.25% as much as 20 ml is then injected into the field.
7. After the needle injection is removed, a block is performed with the same procedure on the opposite side.
8. Evaluation of the success of the M-TAPA block is carried out and monitor the occurrence of blood vessel puncture, hypotension, desaturation, and bradycardia.
9. If hypotension occurs, if the pulse rate is ≥ 60 x / minute, bolus phenylephrine 50 mcg, if the pulse rate is > 60 x / minute, bolus ephedrine 4 mg IV until the mean arterial pressure (MAP) returns to the baseline value. If there is no improvement, it can be repeated at 5-minute intervals. If hypotension persists, norepinephrine is given by titration at a dose of 0.1 mcg / kgBW / minute.
10. If bradycardia occurs with unstable hemodynamics, the patient is given an intravenous injection of atropine sulfate 0.5 mg.
11. If desaturation occurs, perform a physical examination for signs of pneumothorax (lung sounds disappear, hyperresonant percussion), if tension pneumothorax occurs, perform needle decompression then consult a colleague in cardiovascular thoracic surgery (BTKV) for further management.

Group P2 No block is performed, after the operation is completed, extubation preparation is carried out immediately.

Procedures P1 and P2 after surgery:

1. After the block is completed, the patient is given an injection of neostigmine and atropine sulfate to antagonize the remaining atracurium drug still in the patient's body. The patient is extubated after the patient's breathing is adequate and the airway is clear.
2. The patient is observed in the recovery room for 2 hours and transferred to the room if there are no complaints and the Aldrete score is ;9. The pain scale using Numeric Rating Scale is evaluated for the first 0 hours in the recovery room. Observations in the recovery room include: patient complaints, blood pressure, pulse, ECG, respiratory rate and peripheral saturation are carried out every 15 minutes until the patient is transferred to the room. The observation results are recorded on the patient's anesthesia record sheet.
3. After the patient moves to the room, the acute pain service (APS) team will evaluate the pain scale with Numeric Rating Scale (NRS) at 2, 12, 24 hours postoperatively and the total opioid consumption data on the PCA machine will be recorded.
4. Quality of Recovery will evaluate again 24 hours Post Operative.

ELIGIBILITY:
Inclusion Criteria:

1. Patient 18-65 yeasr old
2. IMT 17.5-30 kg/m2
3. Patient with ASA I-II

Exclusion Criteria:

1. Patient Refusal
2. Local Infection
3. Chronic Analgesia drug user

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2024-11-12 (Estimated); Study Completion 2024-11-13 (Estimated)

PRIMARY OUTCOMES:
Proving the effectiveness of postoperative analgesia with Modified-Thoracoabdominal Nerve Block Perichondrial Approach (M-TAPA) in laparoscopic cholecystectomy patients at Prof. I.G.N.G. Ngoerah General Hospital. | 24 hours
  Evaluate total PCA Intravena opioid consumption (morphin in mg) delivered dose.

SECONDARY OUTCOMES:
Numeric rating Scale | 24 hours
  Evaluate Pain Scale using Numeric Rating Scale (NRS) rest and movement 0,2, 12, 24 hours for operative. Range 0-10, 0 is no pain, 10 is severe pain
QoR 40 | 24 hours
  Collect completed questionnaires QoR40 by participant. The score range from 40(Extremely poor quality) to 200 (excellent quality)

CONTACTS AND LOCATIONS:
Overall Officials: WHO WHO, Principal Investigator — World Health Organization
Locations (1):
- Prof I.G.N.G Ngoerah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blythe J, Herrmann E, Faust D, Falk S, Edwards-Lehr T, Stockhausen F, Hanisch E, Buia A. Acute cholecystitis - a cohort study in a real-world clinical setting (REWO study, NCT02796443). Pragmat Obs Res. 2018 Oct 25;9:69-75. doi: 10.2147/POR.S169255. eCollection 2018. PMID 30498388
- [Background] Castillo-Davila LF, Torres-Anaya CJ, Vazquez-Apodaca R, Borboa-Olivares H, Espino-Y-Sosa S, Torres-Torres J. Modified thoracoabdominal nerve block via perichondral approach: an alternative for perioperative pain management in laparoscopic cholecystectomy in a middle-income country. BMC Anesthesiol. 2024 Aug 31;24(1):304. doi: 10.1186/s12871-024-02690-8. PMID 39217281
- [Background] El-Boghdadly K, Pawa A, Chin KJ. Local anesthetic systemic toxicity: current perspectives. Local Reg Anesth. 2018 Aug 8;11:35-44. doi: 10.2147/LRA.S154512. eCollection 2018. PMID 30122981
- [Background] Erbabacan E, Kendigelen P, Koksal GM, Tutuncu C, Ekici BB, Seker TB, Kaya G, Altindas F. Comparison of Transversus Abdominis Plane Block and IV Patient-Controlled Analgesia after Lower Abdominal Surgery. Turk J Anaesthesiol Reanim. 2015 Feb;43(1):24-8. doi: 10.5152/TJAR.2014.82788. Epub 2014 Dec 9. PMID 27366460
- [Background] Fakhoury HMA, Yousef Z, Tamim H, Daher S, Attasi AA, Al Ajlan A, Hajeer AH. Combined effect of age and body mass index on postoperative mortality and morbidity in laparoscopic cholecystectomy patients. Front Surg. 2023 Nov 23;10:1243915. doi: 10.3389/fsurg.2023.1243915. eCollection 2023. PMID 38074287
- [Background] Gungor H, Ciftci B, Alver S, Golboyu BE, Ozdenkaya Y, Tulgar S. Modified thoracoabdominal nerve block through perichondrial approach (M-TAPA) vs local infiltration for pain management after laparoscopic cholecystectomy surgery: a randomized study. J Anesth. 2023 Apr;37(2):254-260. doi: 10.1007/s00540-022-03158-0. Epub 2022 Dec 28. PMID 36575362
- [Background] Tulgar S, Selvi O, Thomas DT, Deveci U, Ozer Z. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides effective analgesia in abdominal surgery and is a choice for opioid sparing anesthesia. J Clin Anesth. 2019 Aug;55:109. doi: 10.1016/j.jclinane.2019.01.003. Epub 2019 Jan 9. No abstract available. PMID 30639940
- [Result] Bilge A, Basaran B, Et T, Korkusuz M, Yarimoglu R, Toprak H, Kumru N. Ultrasound-guided bilateral modified-thoracoabdominal nerve block through a perichondrial approach (M-TAPA) in patients undergoing laparoscopic cholecystectomy: a randomized double-blind controlled trial. BMC Anesthesiol. 2022 Oct 28;22(1):329. doi: 10.1186/s12871-022-01866-4. PMID 36307755
- [Result] Erten E, Kara U, Simsek F, Oztas M, Suzer MA, Kamburoglu H, Eskin MB, Senkal S, Cosar A. Modified thoracoabdominal nerves block through perichondrial approach for laparoscopic cholecystectomy. Rev Assoc Med Bras (1992). 2024 Apr 22;70(3):e20230962. doi: 10.1590/1806-9282.20230962. eCollection 2024. PMID 38655995

DOCUMENTS (1):
  • Informed Consent Form (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT06652581/ICF_000.pdf